CLINICAL TRIAL: NCT00792662
Title: Improving Function, Quality of Life, Glycemia in Diabetics With Dementia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No Subjects enrolled
Sponsor: University of Nebraska (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0470-08-FB
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus; Alzheimer's Disease; Apathy; Dementia
Keywords: Diabetes Mellitus; Alzheimer's Disease; Apathy; Methylphenidate; Dementia
MeSH Terms: conditions — Diabetes Mellitus; Alzheimer Disease; Lethargy; Dementia | interventions — Methylphenidate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): Subject will receive 5mg BID for the first two weeks then 10mg BID until week 16 of the study.
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Standard inactive pill.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Subject will receive 5mg BID for the first two weeks then 10mg BID until week 16 of the study.
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Placebo — Standard inactive pill.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine if the study medication Methylphenidate (Ritalin) will improve subject's blood-sugar control by improving their motivation more than placebo. The secondary objectives of the study are to determine if daily functioning and quality of life improves with methylphenidate treatment.

DETAILED DESCRIPTION:
A total of 50 subjects will be enrolled in this study. This study is being conducted at two sites, UNMC and the Omaha VA Medical Center.

The subject will be asked to take the study drug in the form of a capsule to be taken twice daily. Whether the subject receives methylphenidate or placebo (a pill that has a similar appearance to the study drug, but has no medicine) will be determined by random chance. The probability that the subject will receive methylphenidate is 1 in every 2 subjects or 50% of the time. Subjects receiving methylphenidate will be starting at 5 milligrams (mg) twice daily. Dosage will then be increased to 10mg twice daily at 2 weeks.

After the initial visits, the subjects will be asked to come for follow-up every month for the next 4 visits (sixteen weeks total). During each visit subjects will again be asked questions to assess their motivation, memory, functional status and quality of life. Blood will be drawn and an electrocardiogram (ecg/ekg) will be taken to assess the patient's safety twice during the study.

Partial Compensation may be available for participation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of dementia of the Alzheimer type (Diagnostic and Statistical Manual-IV Text Revision (DSM-IV TR) criteria)
2. Diagnoses of diabetes mellitus type II
3. Poor glycemic control (Hemoglobin A1c (HbA1c ≥ 7.0%))
4. Mild to Moderate Alzheimer's dementia (Mini Mental State Examination (MMSE) >18, but <29)
5. Apathy Evaluation Scale (AES) score of more than 30
6. Ability to provide informed consent by either the patient or caregiver.
7. If subjects are being treated with antidepressants, they should be on a stable dose of antidepressants for at least two months prior to the enrollment into the study.
8. If subjects are being treated with cholinesterase inhibitors and memantine, they should be on stable dose of those medications at least four months prior to the enrollment into the study.
9. Subjects should be on stable dose of statins and ACE inhibitors for ≥ 2 months.
10. Subjects should be on stable dose of diabetes treatment for 2 months prior to enrollment.

Exclusion Criteria:

1. Severe dementia (MMSE < 18)
2. Patient currently taking methylphenidate or hypersensitivity or prior significant adverse events with methylphenidate.
3. Patients currently taking Adderall (amphetamine mixed salts) or Dexedrine (dextroamphetamine sulphate) or any other amphetamine product.
4. Uncontrolled hypertension (BP > 140/90) or tachycardia (100) at screening visit
5. Patients with frontotemporal dementia
6. Patients meeting criteria for Major Depressive Disorder on the Mini International Neuropsychiatric Inventory (MINI)
7. Patients with active psychosis as determined by MINI
8. Patients currently being treated with antipsychotics
9. History of uncontrolled seizure disorder
10. History of malignant hypertension, symptomatic cardiovascular disease, cardiomyopathy, known structural cardiac defect or medically unstable arrhythmias.
11. History of Tourette's syndrome or presence of motor tics
12. Patients with glaucoma
13. Patients taking monoamine oxidase inhibitors (MAOIs)
14. Patient taking clonidine
15. Patients being treated with insulin pump

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11-18 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2011-12-20 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C as a Marker for Glycemic Control | 16 weeks
  Hemoglobin A1C (HbA1c) will be used as marker for glycemic control. It is accepted as the best marker for glycemic control in the previous 120 days. Changes in HbA1c are clinically meaningful.

SECONDARY OUTCOMES:
Apathy Evaluation Scale-Clinician (AES-C) | 16 weeks
  Apathy Evaluation Scale-Clinician (AES-C): The clinician-rated version will be used for this project. This 18 item scale with scores ranging from 18 to 72, assesses apathy in behavioral, cognitive and emotional domains over the previous four weeks.
Clinical Global Impression (CGI) Scale | 16 weeks
  Clinical Global Impression (CGI): This is an observational scale of global evaluation with two components-the CGI-Severity, which rates illness severity (1=normal, not at all ill to 7=among the most extremely ill patients) and the CGI-Improvement, which rates change from the initiation (baseline) of treatment (1=very much improved since the initiation of treatment to 7=very much worse since the initiation of treatment.")
Instrumental Activities of Daily Living (IADL) Scale | 16 weeks
  Instrumental Activities of Daily Living (IADL): It is a survey assessing eight domains of higher functions necessary to live independently. It is rated from 0 (low functioning) to 23 (high functioning) based on the independent living of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad R Padala, M.D., Principal Investigator — University of Nebraska